CLINICAL TRIAL: NCT05354180
Title: Comparison of Navicular Mobilization and Rigid Tape in Pes Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC -01256 Samra Ismail
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Pes Planus
Keywords: pain; navicular mobilization; rigid tape; tibial torsion
MeSH Terms: conditions — Flatfoot; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- navicular mobilization (Experimental): Plantar glide combined with rotation of navicular bone against the talus The glide will be given in 20 repetitions of 3 sets, for 5 days a week
  Interventions: Other: navicular mobilization
- rigid tapping (Experimental): A non-elastic zinc oxide sports tape will be applied to patients. Patient will be advised to protect the tape from getting wet.
  Tape will be changed on every 3rd day (48 hours) on Wednesday and Friday.
  Interventions: Other: rigid tapping
- Navicular Mobilization and Rigid Taping| (Experimental): Plantar glide combined with rotation of navicular bone against the talus The glide will be given in 20 repetitions of 3 sets, for 5 days a week.
  A non-elastic zinc oxide sports tape will be applied to patients. Patient will be advised to protect the tape from getting wet.
  Tape will be changed on every 3rd day (48 hours) on Wednesday and Friday.
  Interventions: Other: Navicular Mobilization and Rigid Taping

INTERVENTIONS:
Other: navicular mobilization — Plantar glide combined with rotation of navicular bone against the talus The glide will be given in 20 repetitions of 3 sets, for 5 days a week
  Arms: navicular mobilization
Other: rigid tapping — A non-elastic zinc oxide sports tape will be applied to patients. Patient will be advised to protect the tape from getting wet.
  Tape will be changed on every 3rd day (48 hours) on Wednesday and Friday.
  Arms: rigid tapping
Other: Navicular Mobilization and Rigid Taping — Plantar glide combined with rotation of navicular bone against the talus The glide will be given in 20 repetitions of 3 sets, for 5 days a week.
  A non-elastic zinc oxide sports tape will be applied to patients. Patient will be advised to protect the tape from getting wet.
  Tape will be changed on every 3rd day (48 hours) on Wednesday and Friday.
  Arms: Navicular Mobilization and Rigid Taping|

SUMMARY:
Pes planus, sometimes known as flat feet, is one of these disorders and is characterized by a collapsed medial longitudinal arch, hindfoot eversion, and forefoot abduction. Pes planus is a musculoskeletal condition that causes hip, knee, and foot discomfort. According to a descriptive cross-sectional survey, 17% of school-aged children, 64% men and 34% females have flat foot deformity. Talonavicular joint is responsible for translating inversion and eversion movements of the foot. Mobilization of the Talonavicular joint helps in the improvement of joint dysfunction caused by inappropriate or bad posture via the proprioceptors.

Rigid tape also known as low dye tape is defined as non-elastic zinc oxide tape used by physical therapists to stabilize a joint and limit movement. The conventional rigid tape is frequently used with non-contractile tissue, which then acts similarly to a ligament to limit joint mobility and prevent joints from moving into dangerous or end range positions.

DETAILED DESCRIPTION:
Foot disorders are very frequent in elder adults, with some illnesses having a prevalence of up to 65 percent. Foot diseases and accompanying symptoms have been linked to a variety of negative health outcomes, including falls and functional restrictions. The biomechanics of many foot problems, however, are yet unknown. Foot biomechanics during functional activities, such as walking could play a role in the onset and progression of foot problems.

Pes planus, sometimes known as flat feet, is one of these disorders and is characterized by a collapsed medial longitudinal arch, hindfoot eversion, and forefoot abduction. Pes planus is a musculoskeletal condition that causes hip, knee, and foot discomfort.

Pes planus is a common deformity that affects newborns and children and normally goes away by the time they reach puberty. After that, the incidence tends to drop with age, with just 4% of children having flatfoot by the age of ten. This backs up the assumption that flatfoot in children normally resolves on its own throughout the first ten years of life.

Pes planus is divided into two types: flexible (functional) and rigid (structural).

The initial treatment of painful-but-flexible flatfoot is nonoperative. Conservative therapy techniques such as rest, icing, massage, and nonsteroidal anti inflammatory medication, should always be used initially to reduce pain in symptomatic flexible and rigid flatfeet. Physical therapy plan which includes electrotherapy, Achilles' tendon stretching , strengthening of calf muscles, intrinsic muscles of the foot, and navicular mobilization are used as treatment options.

Talo-navicular joint is responsible for translating inversion and eversion movements of the foot. Mobilization of the talo-navicular joint helps in the improvement of joint dysfunction caused by inappropriate or bad posture via the proprioceptors.

Rigid tape also known as low dye tape(18) is defined as non-elastic zinc oxide tape used by physical therapists to stabilize a joint and limit movement. The conventional rigid tape is frequently used with non-contractile tissue, which then acts similarly to a ligament to limit joint mobility and prevent joints from moving into dangerous or end range positions.

ELIGIBILITY:
Inclusion Criteria:

* Children with neuromuscular disorders level I, II and III according to gross motor function classification system
* Positive Navicular Drop (navicular drop test) less than ≥ 10 mm

Exclusion Criteria:

* Other deformities of foot.
* Overweight and obesity.
* Any recent lower limb injury in past 6 months.
* Any fracture in last 6 months.
* Taken any pain killer injection..
* Any recent lower limb surgery in past 6 months.
* Myopathies

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
Numerical pain rating scale | four weeks
  a 11 point outcome measure used to measure the intensity of pain ranging from 0 (no pain) to 10 (worst imaginable pain(23), it has been exhibited moderate reliability (Intra class correlation coefficient (ICC) is a widely used reliability index) is 0.67. Assessment to be done at baseline and at end of every week.
Time up & go test. | four weeks
  used to asses functional mobility and balance in which subject rise from a chair, walk 3 meter or 10 feet , turn around, return to the chair, and sit down.the performance is graded based on whether the individual completes the test under 10 sec(independent), under 20 sec(independent for main transfers) and under 30 sec (require assistance).It has good to excellent reliability results with intraclass correlation coefficients ICC range,0.69-.99.Assessment to be done at baseline and at end of every week.
Goniometer | four weeks
  (tool used by health professionals to objectively measure the range of motion of each joint effectively). The data analysis demonstrated that the goniometer has high intertester reliability with ICC ranges from 0.98-0.99.
  Assessment to be done at baseline and at end of every week.
Navicular drop test | four weeks
  The navicular drop test is a measure to evaluate the function of the medial longitudinal arch, which is important for examination of patients with overuse injuries It evaluates the foot hyper pronation by first measuring the navicular tuberosity height from floor or supporting surface in seated position and then in full weight bearing position by placing an index card at medial aspect of foot and then measuring the difference between the two marks of navicular level in millimeters. This procedure was performed bilaterally and navicular drop values greater than 10 mm are considered to be hyper pronation(22).It has high intraclass correlation coefficients reported for both intertester and intratester reliability ranging from 0.78 to 0.83.
  Assessment to be done at baseline and at end of every week.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Zobia School for special children, Mirpur, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No